CLINICAL TRIAL: NCT05541653
Title: A Randomized Controlled Trial of Concentrated Investment in Black Neighborhoods to Address Structural Racism as a Fundamental Cause of Poor Health
Brief Title: The IGNITE Study on Concentrated Investment in Black Neighborhoods
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Eugenia Garvin, Assistant Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 850178
Record Dates: First submitted 2022-09-02; First posted 2022-09-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Financial Stress; Economic Problems; Environmental Exposure; Health Behavior; Health, Subjective; Mental Health Wellness 1
MeSH Terms: conditions — Financial Stress; Health Behavior

STUDY DESIGN:
Masking Description: The investigators are not masked. Our recruitment team will be masked until cluster recruitment is complete. The outcomes assessor will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): At the individual level, participants in the intervention arm receive place-based and financial well-being interventions.
  These include, at the individual level:
  * Tax preparation
  * Access to public benefits
  * Financial counseling and microgrants
  At the neighborhood level:
  * Abandoned house remediation
  * Trash cleanup
  * Vacant lot greening
  * Tree planting
  Interventions: Other: Financial Well-being Interventions; Other: Place-based Interventions
- Control (No Intervention): Participants in the control arm will not receive any of the listed interventions.

INTERVENTIONS:
Other: Financial Well-being Interventions — Tax preparation; access to public benefits; financial counseling and microgrants
  Arms: Intervention
Other: Place-based Interventions — Vacant lot greening; abandoned house remediation; trash cleanup; and tree planting.
  Arms: Intervention

SUMMARY:
Black Americans in the US fare worse across nearly every health indicator compared to White individuals. In Philadelphia, the location of this study, these health disparities culminate in a stark longevity gap, with average life expectancies in poor, predominantly Black neighborhoods being 20 years lower than in nearby affluent, predominantly White neighborhoods. The investigators will conduct a cluster randomized controlled trial (RCT) of a suite of place-based and financial-wellbeing interventions at the community, organization, and individual/household levels that address the social determinants of racial health disparities. At the community level, the investigators address underinvestment in Black neighborhoods by implementing vacant lot greening, abandoned house remediation, tree planting, and trash cleanup. At the organization level, the investigators partner with community-based financial empowerment providers to develop cross-organizational infrastructure to increase reach and maximize efficiency. At the individual/household levels, the investigators increase access to public benefits, financial counseling and tax preparation services, and emergency cash assistance. The investigators will test this "big push" intervention in 60 Black neighborhood microclusters, with a total of 720 adults. The investigators hypothesize that this "big push" intervention will have significant impact on overall health and wellbeing.

DETAILED DESCRIPTION:
Black individuals in the United States fare worse than White individuals across almost every social, economic, and health indicator. The Black health disadvantage starts at birth, reflecting the cumulative toll of racialized social stressors and healthcare discrimination on maternal health and resulting in higher rates of preterm birth and low birth weight. Black youth are disproportionately exposed to environmental toxins such as lead and adverse childhood events such as financial hardship and neighborhood violence. Black adults have higher rates of chronic disease, including diabetes, hypertension, as well as many cancers. These and other forces culminate in a stark racial longevity gap: in Philadelphia, the location of this study, life expectancy for people living in a poor, predominantly Black neighborhood is 20 years lower than for people living in a nearby affluent, predominantly White neighborhood.

The fundamental cause of these striking and pervasive disparities is structural racism - the confluence of deep historical, institutional, cultural, and ideological forces that unequally distribute resources and risks across racialized groups. Structural racism patterns health by affecting a range of interconnected, mutually reinforcing social determinants of health at the national, neighborhood, household, and individual levels. Most notably, longstanding, systematic disinvestment has resulted in highly segregated Black neighborhoods with dilapidated environmental conditions and severe economic insecurity within Black households, leading to a "feedback loop of concentrated racial disadvantage," all of which have been strongly tied to poor health.

Most interventions seeking to address racial health disparities focus on individual-level behaviors and outcomes, or individual channels by which structural racism harms health. However, by failing to address upstream social determinants, these interventions have had limited population level impact. A multi-level, multi-component intervention package focused on a range of social determinants of health is necessary to meaningfully address structural racism as a fundamental cause of racial health disparities.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Have the ability to communicate via text messaging
* Individuals comfortable communicating in English
* A permanent resident of the home where they are to be enrolled
* Have knowledge of their household finances

Exclusion Criteria:

* Individuals who plan to move out of the study microcluster within 6 months
* Individuals who are unable to fully consent and participate based on recruitment team assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Health Index | 24 months
  Composite index using method of Anderson (2008) based on three questions: rating of overall health (5-pt Likert ranging from poor to excellent); rating of how health has changed in last 6 months (better, same, worse); and number of days in the last 30 where physical or mental health precluded engagement in usual activities (self-care, work, recreation); (Oregon Health Insurance Experiment)
Psychological Distress | 24 months
  Kessler-6 (answers scored 0-24 with higher scores indicating higher levels of psychological distress)

SECONDARY OUTCOMES:
Overall health | 24 months
  Rating of overall health (5-pt Likert ranging from poor to excellent) (Oregon Health Insurance Experiment)
Poor health | 24 months
  Whether individual reported either poor or fair health to overall health question (Oregon Health Insurance Experiment)
Change in overall health | 24 months
  Rating of how health has changed in last 6 months (better, same, worse)
Healthy days | 24 months
  Number of days in the last 30 where physical or mental health precluded engagement in usual activities (self-care, work, recreation)
Sleep duration | 24 months
  Number of hours of usual sleep (Behavioral Risk Factor Surveillance System)
Short sleep | 24 months
  Less than seven hours of usual night sleep (Behavioral Risk Factor Surveillance System)
Healthcare access | 24 months
  Received all needed care in the last 6 months (Behavioral Risk Factor Surveillance System)
Financial well-being | 24 months
  Consumer Financial Protection Bureau, Abbreviated Financial Well-being Survey
Food insecurity | 24 months
  Current Population Survey Food Security Supplement Screener
Income tax filing | 24 months
  Whether or not individual (or someone in household on behalf of individual) filed previous years income tax (yes, planning to file late, no) (internally developed)
Home ownership | 24 months
  Whether or not individual owns house, condo, or mobile home (Add Health)
Owing on mortgage | 24 months
  Whether or not individual has remaining mortgage payments (internally developed)
Total debt | 24 months
  Amount of debt added altogether, not including mortgage (Add Health)
Participation in public medical benefit programs | 24 months
  Participation of a household member (including respondent) in Medicaid, Medicare, Medicare savings, LIS, CHIP, Qualified Health Plans, SelectPlan, other, or none (internally developed)
Participation in public food benefit programs | 24 months
  Participation of a household member (including respondent) in SNAP, WIC, Senior Food Box, other, or none (internally developed)
Participation in public income support or cash benefit programs | 24 months
  Participation of a household member (including respondent) in TANF, LIHEAP, SSI/SSDI, UI, PA General Assistance, PA Emergency Rental Assistance, EITC, CTC Refugee Cash Assistance, CCIS, PA Child Care Tax Credit, other, or none (internally developed)
Participation in public home ownership benefit programs | 24 months
  Participation of a household member (including respondent) in PTRR, Homestead Exemption, LOOP, Basic Systems Repair Program, PA Homeowner Assistance, Philly First Home Program, Philadelphia Home Repair Assistance, other or none (internally developed)
Frequency of greenspace engagment | 24 months
  Frequency with which individual visits a greenspace (such as a park, garden, greened vacant lot, trail, or any other outdoor space with vegetation) (adapted from Evenson et al 2013 Environment and Behavior)
Time spent in greenspace | 24 months
  Time spent in a greenspace on a typical day (adapted from Evenson et al 2013 Environment and Behavior))
Reasons for not spending time in greenspace | 24 months
  Things that stop an individual from spending time in greenspace (adapted from Evenson et al 2013 Environment and Behavior)
Perception of tree cover | 24 months
  Beliefs about number of trees in the neighborhood (internally developed)
Tree planting concerns | 24 months
  Whether or not individual has concerns about planting more trees in neighborhood (internally developed)
Perceived tree health benefits | 24 months
  Whether or not individual believes trees confer health benefits (e.g., safety, mental health benefits, physical health benefits, social benefits, environmental benefits, aesthetic benefits)
Perceived stress | 24 months
  Perceived Stress Scale (responses scored 0-16 with higher scores correlated to higher stress)
Time spent in neighborhood | 24 months
  Frequency with which individual endorses spending time relaxing, socializing, or hanging out in porches, stoops, and front yards of neighborhoods (adapted from Kahneman et al 2004 Science)
Neighborhood social capital | 24 months
  Neighborhood Social Cohesion & Exchange and Social & Physical Disorder Scale (two domains: Social Cohesion and Physical Disorder. Higher scores for social cohesion indicate higher levels of social cohesion and higher scores for physical disorder indicate higher levels of physical disorder).
Physical disorder | 24 months
  Whether or not participant reports a lot of abandoned buildings in their neighborhood (Ross and Mirowksi)
Neighborhood crime rates | Quarterly data from 24 months (8 quarters) prior to enrollment and 12 months (4 quarters) after intervention period complete
  Overall number of crimes, number of violent crimes, serious crimes, and gun related incidents
Nuisance calls | Quarterly data from 24 months (8 quarters) prior to enrollment and 12 months (4 quarters) after intervention period complete
  Number of 311 calls and number of 311 calls for neighborhood cleanup and remediation-related issues

CONTACTS AND LOCATIONS:
Locations (1):
- Philadelphia Neighborhoods, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT05541653/Prot_002.pdf
  • Statistical Analysis Plan (2026-02-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT05541653/SAP_003.pdf